CLINICAL TRIAL: NCT02366728
Title: Evaluation of Overcoming Limited Migration and Enhancing Cytomegalovirus-specific Dendritic Cell Vaccines With Adjuvant TEtanus Pre-conditioning in Patients With Newly-diagnosed Glioblastoma
Brief Title: DC Migration Study for Newly-Diagnosed GBM
Acronym: ELEVATE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mustafa Khasraw, MBChB, MD, FRCP, FRACP (Other)
Responsible Party: Sponsor-Investigator, Mustafa Khasraw, MBChB, MD, FRCP, FRACP, Professor, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00054740
Record Dates: First submitted 2014-10-28; First posted 2015-02-19 (Estimated); Results first posted 2022-02-01 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Glioblastoma; Astrocytoma, Grade IV; Giant Cell Glioblastoma; Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide; Sodium Chloride; Basiliximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group I: Unpulsed DC pre-conditioning (Experimental): 0.4 mLs of 1 x 10^6 autologous unpulsed DCs in saline will be administered to a single side of the groin, and 0.4 mLs of saline administered to the contralateral side 1 day prior to the 4th human CMV pp65-LAMP mRNA-pulsed autologous DCs vaccine. pp65 DC Vaccine #4 is 111In-labeled DCs for migration studies.
  Interventions: Biological: Unpulsed DCs; Biological: Human CMV pp65-LAMP mRNA-pulsed autologous DCs; Biological: 111In-labeled DCs; Drug: Temozolomide; Drug: Saline
- Group II: Tetanus pre-conditioning (Experimental): Tetanus diptheria toxoid (Td) (1 flocculation unit) will be administered to a single side of the groin, and 0.4 mLs of saline administered to the contralateral side 1 day prior to the 4th human CMV pp65-LAMP mRNA-pulsed autologous DCs vaccine. pp65 DC Vaccine #4 is 111In-labeled DCs for migration studies.
  Interventions: Biological: Td; Biological: Human CMV pp65-LAMP mRNA-pulsed autologous DCs; Biological: 111In-labeled DCs; Drug: Temozolomide; Drug: Saline
- Group III: Basiliximab and Tetanus pre-conditioning (Experimental): Basiliximab infusions prior to human CMV pp65-LAMP mRNA-pulsed autologous DCs vaccines #1 and #2 with Td pre-conditioning (1 flocculation unit) will be administered to a single side of the groin, and 0.4 mLs of saline administered to the contralateral side 1 day prior to the 4th human CMV pp65-LAMP mRNA-pulsed autologous DCs vaccine.
  Interventions: Biological: Human CMV pp65-LAMP mRNA-pulsed autologous DCs; Drug: Temozolomide; Drug: Saline; Drug: Basiliximab

INTERVENTIONS:
Biological: Unpulsed DCs — Patients in Group I will receive 1 x 10^6 autologous unpulsed DCs in saline administered to a single side of the groin intradermally 1 day before the fourth vaccine.
  Other Names: Unpulsed DCs pre-conditioning
  Arms: Group I: Unpulsed DC pre-conditioning
Biological: Td — Patients in Groups II and III will receive a single dose of Td toxoid (1 flocculation unit, Lf, in 0.4 mLs) administered to a single side of the groin given intradermally 1 day before the fourth vaccine.
  Other Names: Td toxoid; Td pre-conditioning
  Arms: Group II: Tetanus pre-conditioning
Biological: Human CMV pp65-LAMP mRNA-pulsed autologous DCs — 2x10^7 human CMV pp65-LAMP mRNA-pulsed autologous DCs are given intradermally and bilaterally at the groin site (divided equally to both inguinal regions). Patients will receive up to a total of 10 DC vaccines.
  Other Names: CMV-specific dendritic cell vaccine; DCs
Biological: 111In-labeled DCs — 111In-labeled DCs are 2 x 10^7 pp65-LAMP mRNA loaded mature DCs will be labeled with 111In (50 μCi / 5 x 10^7 DCs) and given i.d. as fourth vaccine for Groups I and II only.
  Arms: Group I: Unpulsed DC pre-conditioning; Group II: Tetanus pre-conditioning
Drug: Temozolomide — Temozolomide is a standard chemotherapy given to all enrolled patients at a targeted dose of 150-200mg/m2/d for 5 days every 5 (± 1) weeks for a total of 6 to 12 cycles at the discretion of the treating oncologist.
  Other Names: Temodar; TMZ
Drug: Saline — 0.4mL of saline given in the opposite groin 1 day before the fourth vaccine in all groups
Drug: Basiliximab — Group III will receive basiliximab infusions (20 mg I.V) 1 week before the first vaccine and 1 week before the second vaccine.
  Arms: Group III: Basiliximab and Tetanus pre-conditioning

SUMMARY:
This randomized phase II study will assess the impact of pre-conditioning on migration and survival among newly diagnosed glioblastoma (GBM) patients who have undergone definitive resection and completed standard temozolomide (TMZ) and radiation treatment, as well as the impact of tetanus pre-conditioning and basiliximab together on survival. After completing standard of care radiotherapy with concurrent TMZ, patients will be randomized to 1 of 3 treatment arms: 1). receive cytomegalovirus (CMV)-specific dendritic cell (DC) vaccines with unpulsed (not loaded) DC pre-conditioning prior to the 4th vaccine; 2). receive CMV-specific DC vaccines with Tetanus-Diphtheria Toxoid (Td) pre-conditioning prior to the 4th vaccine; 3). receive basiliximab infusions prior to the 1st and 2nd DC vaccines along with Td pre-conditioning prior to the 4th vaccine. A permuted block randomization algorithm using a 1:1:1 allocation ratio will be used to assign patients to a treatment arm. Randomization will be stratified by CMV status (positive, negative), with the assignment to arms I and II being double-blinded. Effective March 2017, randomization to Group III has been terminated.

DETAILED DESCRIPTION:
A maximum of 100 patients with resected, newly-diagnosed World Health Organization (WHO) Grade IV GBM will be enrolled in this study with the expectation that approximately 79 patients will be randomized to subsequent treatment after completion of radiation treatment with concurrent temozolomide. Effective March 2017, randomization to Group III has been terminated. All consented patients will undergo a leukapheresis after resection for harvest of Peripheral Blood Lymphocytes (PBLs) for generation of DCs. Patients will then receive Radiation Therapy (RT) and concurrent TMZ at a standard targeted dose of 75 mg/m^2/d. Patients should start RT within approximately 6 weeks of surgery. Patients who experience progressive disease during radiation, are dependent on steroid supplements above physiologic levels at time of first vaccination, are unable to tolerate TMZ, or whose DCs or PBLs fail to meet release criteria will be withdrawn from the study and replaced and will not undergo repeat leukapheresis. For patients whose initial leukapheresis yields less than 3 vaccines, repeat leukapheresis may be obtained a minimum of 2 weeks from the previous leukapheresis (and may be repeated as needed) if pre-pheresis blood work is within the Apheresis Center's parameters and as long as this does not cause a significant delay in treatment for the patient.

After RT and concurrent TMZ, patients will then be randomized and begin the initial cycle of TMZ at a standard targeted dose of 150-200mg/m^2/d for 5 days at the discretion of the treating oncologist 4 (± 2) weeks after completing RT. The study cycle of TMZ comprises a targeted dose of 150-200mg/m^2/d for 5 days every 5 (± 1) weeks. All patients will receive up to a total of 10 DC vaccines given bilaterally at the groin site unless progression occurs. DC vaccines will be given intradermally (i.d.) and divided equally to both inguinal regions. DC vaccines #1-3 will be given every two weeks, thus delaying the initiation of TMZ cycle 2. Patients will then be vaccinated in conjunction with subsequent TMZ cycles every 5 (± 1) weeks for a total of 6 to 12 cycles after RT at the discretion of the treating oncologist. DCs will be given on day 21 ± 2 days of each TMZ cycle. DC vaccinations will continue during TMZ cycles up to a total of 10 unless progression occurs.

Before the first DC vaccination, all patients will receive immunization with 0.5 mL of Td intramuscularly into the deltoid muscle to ensure adequate immunity to the tetanus antigen. Those assigned to Group III will receive basiliximab 20 mg infusions 1 week before the 1st and 1 week before the 2nd vaccine. At the time of the fourth DC vaccine, patients will receive pre-conditioning per the assigned group (Group I-unpulsed DCs i.d.; Group II- Td i.d.; Group III-Td i.d.). A single dose of Td toxoid (1 flocculation unit, in 0.3 milliliters (mLs) of saline for a total volume of 0.4 mLs) or 0.4 mLs of 1 x 10^6 autologous unpulsed DCs in saline will be administered to a single side of the groin, and 0.4 mLs of saline administered to the contralateral side 12-24 hours prior to the fourth DC vaccine, which is always given bilaterally at the groin site. Patients in Groups I and II will then receive 111In-labeled DCs to compare the effects of different skin preparations on DC migration followed by Single-Photon Emission Computed Tomography and Computed Tomography (SPECT/CT) imaging immediately and at 1 and 2 days after injection. Group III will not undergo migration studies. Groups I and II will be double blinded. Group III will not be blinded.

All patients will undergo leukapheresis again for immunologic monitoring with specific assessment of baseline antigen-specific cellular and humoral immune responses and further DC generations 4 (± 2) weeks after vaccine #3. Patients will be imaged bimonthly without receiving any other prescribed anti-tumor therapy. Patients will undergo an additional leukapheresis for generation of DCs if needed to continue vaccinations.

As part of standard care for these patients, upon tumor progression, participants may undergo stereotactic biopsy or resection. As this is not a research procedure consent will be obtained separately. However, if tissue is obtained, it will be used to confirm tumor progression histologically and to assess immunologic cell infiltration and pp65 antigen escape at the tumor site.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years of age
* WHO Grade IV Glioma with definitive resection prior to enrollment, with residual radiographic contrast enhancing disease on the post-operative CT or Magnetic Resonance Imaging (MRI) of <1 cm in maximal diameter in any axial plane
* MRI post radiation therapy (RT) does not show progressive disease at time of randomization
* Karnofsky Performance Status of > 80%.
* Hemoglobin ≥ 9.0 g/dl, Absolute Neutrophil Count ≥ 1,500 cells/µl, platelets ≥ 125,000 cells/µl
* Serum creatinine ≤ 1.5 mg/dl, Serum Glutamic Oxaloacetic Transaminase & bilirubin ≤ 1.5 times upper limit of normal
* Signed informed consent approved by the Institutional Review Board
* Female patients must not be pregnant or breast-feeding. Female patients of childbearing potential (defined as < 2 years after last menstruation or not surgically sterile) must use a highly effective contraceptive method (allowed methods of birth control, [i.e. with a failure rate of < 1% per year] are implants, injectables, combined oral contraceptives, intra-uterine device [IUDs; only hormonal], sexual abstinence or vasectomized partner) during the trial & for a period of > 6 months following the last administration of trial drug(s). Female patients with an intact uterus (unless amenorrhea for the last 24 months) must have negative serum pregnancy test within 48 hours prior to first study procedure (leukapheresis).
* Fertile male patients must agree to use a highly effective contraceptive method (allowed methods of birth control [i.e. with a failure rate of < 1% per year] include a female partner using implants, injectables, combined oral contraceptives, IUDs [only hormonal], sexual abstinence or prior vasectomy) during the trial & for a period of > 6 months following the last administration of trial drugs

Exclusion Criteria:

* Pregnant or breast-feeding
* Women of childbearing potential & men who are sexually active and not willing/able to use medically acceptable forms of contraception
* Patients with known potentially anaphylactic allergic reactions to gadolinium-Diethylenetriaminepentaacetic Acid
* Patients who cannot undergo MRI or SPECT due to obesity or to having certain metal in their bodies (specifically pacemakers, infusion pumps, metal aneurysm clips, metal prostheses, joints, rods, or plates)
* Patients with evidence of tumor in the brainstem, cerebellum, or spinal cord, radiological evidence of multifocal disease, or leptomeningeal disease
* Severe, active comorbidity, including any of the following

  * Unstable angina and/or congestive heart failure requiring hospitalization
  * Transmural myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of study initiation
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy
  * Known hepatic insufficiency resulting in clinical jaundice and/or coagulation defects;
  * Known Human Immunodeficiency Virus positive status
  * Major medical illnesses or psychiatric impairments that, in the investigator's opinion, will prevent administration or completion of protocol therapy
  * Active connective tissue disorders, such as lupus or scleroderma that, in the opinion of the treating physician, may put the patient at high risk for radiation toxicity
* Co-medication that may interfere with study results; e.g. immuno-suppressive agents other than corticosteroids;
* Prior, unrelated malignancy requiring current active treatment with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin;
* Patients are not permitted to have had any other conventional therapeutic intervention other than steroids prior to enrollment outside of standard of care chemotherapy & radiation therapy. Patients who receive previous inguinal lymph node dissection, radiosurgery, brachytherapy, or radiolabeled monoclonal antibodies will be excluded
* Current, recent (within 4 weeks of the administration of this study agent), or planned participation in an experimental drug study
* Known history of autoimmune disease (with the exceptions of medically-controlled hypothyroidism and Type I Diabetes Mellitus)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-10-12 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dina Randazzo, DO, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group I: Unpulsed DC Pre-conditioning | Group II: Tetanus Pre-conditioning | Group III: Basiliximab and Tetanus Pre-conditioning
Started | 27 | 28 | 9
Received at Least One ppp65 Vaccine | 25 | 27 | 8
Completed | 23 | 27 | 8
Not Completed | 4 | 1 | 1
Not completed — Death | 0 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Screen Failure | 2 | 1 | 0
Not completed — Only yielded 2 vaccines | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants who received at least one ppp65 vaccine.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I: Unpulsed DC Pre-conditioning | Group II: Tetanus Pre-conditioning | Group III: Basiliximab and Tetanus Pre-conditioning | Total
Number analyzed (Participants) | 25 | 27 | 8 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (13.3) | 53.7 (13.6) | 50.4 (12.4) | 54.1 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 2 | 18
  Male | 19 | 17 | 6 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 22 | 25 | 7 | 54
  Unknown or Not Reported | 3 | 2 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 23 | 25 | 8 | 56
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 27 | 8 | 60

OUTCOME MEASURES:

1. Primary Outcome: Median Overall Survival
Description: Overall survival will be defined as the time in months between randomization and death, or last follow-up if alive. Kaplan-Meier methods will be used to estimate overall survival.
Time Frame: Up to 72 months (from the time of randomization of the first patient until approximately 31 months after randomization of the last patient)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group I: Unpulsed DC Pre-conditioning | Group II: Tetanus Pre-conditioning | Group III: Basiliximab and Tetanus Pre-conditioning
Number analyzed (Participants) | 25 | 27 | 8
months | 16 [12.8 to 25.5] | 20 [16.7 to 25.6] | 19 [10.26 to NA] — An estimation was not possible due to an insufficient number of participants experiencing events.
Statistical Analysis 1: Comparison: Group I: Unpulsed DC Pre-conditioning vs Group II: Tetanus Pre-conditioning; Test type: Other; p = 0.072, Log Rank
Statistical Analysis 2: Comparison: Group I: Unpulsed DC Pre-conditioning vs Group III: Basiliximab and Tetanus Pre-conditioning; Test type: Other; p = 0.089, Log Rank

2. Primary Outcome: Percentage of 111In-labeled Dendritic Cells Migrating to the Inguinal Lymph Nodes
Description: Within Groups I and II only, the percentage of 111In-labeled DCs migrating to the inguinal lymph nodes from the initial injection sites in the left and right groin at 48 hours post-vaccination #4 will be calculated.
Time Frame: For each patient, migration studies will occur after vaccination #4 which occurs approximately 7 months after study consent.
Population: Data not collected on the Basiliximab and Tetanus pre-conditioning group.
Measure: Median (Inter-Quartile Range); unit: percentage of cells
Arm/Group | Group I: Unpulsed DC Pre-conditioning | Group II: Tetanus Pre-conditioning | Group III: Basiliximab and Tetanus Pre-conditioning
Number analyzed (Participants) | 25 | 27 | 0
percentage of cells | 6.0 [3.0 to 8.0] | 9 [6.5 to 11.0] |
Statistical Analysis 1: Comparison: Group I: Unpulsed DC Pre-conditioning vs Group II: Tetanus Pre-conditioning; Test type: Other; p = 0.0195, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Median Overall Survival in CMV Positive Participants
Description: Median overall survival will be estimated in the subset of participants that are CMV positive. Overall survival will be defined as the time in months between randomization and death, or last follow-up if alive. Kaplan-Meier methods will be used to estimate overall survival.
Time Frame: as for outcome 1
Population: Participants who are CMV positive. Data not collected on the Basiliximab and Tetanus pre-conditioning group.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group I: Unpulsed DC Pre-conditioning | Group II: Tetanus Pre-conditioning | Group III: Basiliximab and Tetanus Pre-conditioning
Number analyzed (Participants) | 9 | 11 | 0
months | 16.5 [12.8 to 44.1] | 23.8 [19.9 to NA] — An estimation was not possible due to an insufficient number of participants experiencing events. |
Statistical Analysis 1: Comparison: Group I: Unpulsed DC Pre-conditioning vs Group II: Tetanus Pre-conditioning; Test type: Other; p = 0.40, Log Rank

4. Primary Outcome: Median Overall Survival in CMV Negative Participants
Description: Median overall survival will be estimated in the subset of participants that are CMV negative. Overall survival will be defined as the time in months between randomization and death, or last follow-up if alive. Kaplan-Meier methods will be used to estimate overall survival.
Time Frame: as for outcome 1
Population: Participants who are CMV negative. Data not collected on the Basiliximab and Tetanus pre-conditioning group.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group I: Unpulsed DC Pre-conditioning | Group II: Tetanus Pre-conditioning | Group III: Basiliximab and Tetanus Pre-conditioning
Number analyzed (Participants) | 16 | 16 | 0
months | 13.4 [9.5 to 26.1] | 16.7 [13.6 to 45.6] |
Statistical Analysis 1: Comparison: Group I: Unpulsed DC Pre-conditioning vs Group II: Tetanus Pre-conditioning; Test type: Other; p = 0.40, Log Rank

5. Secondary Outcome: Median Progression-free Survival
Description: Progression-free survival will be defined as the time in months between randomization and disease progression or death. Participants alive without disease progression will be censored at the time of their last follow-up. Kaplan-Meier methods will be used to estimate progression-free survival.
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group I: Unpulsed DC Pre-conditioning | Group II: Tetanus Pre-conditioning | Group III: Basiliximab and Tetanus Pre-conditioning
Number analyzed (Participants) | 25 | 27 | 8
months | 6.5 [4.4 to 12.1] | 6.7 [4.6 to 15.2] | 7.1 [6.0 to NA] — An estimation was not possible due to an insufficient number of participants experiencing events.
Statistical Analysis 1: Comparison: Group I: Unpulsed DC Pre-conditioning vs Group II: Tetanus Pre-conditioning; Test type: Other; p = 0.16, Log Rank
Statistical Analysis 2: Comparison: Group I: Unpulsed DC Pre-conditioning vs Group III: Basiliximab and Tetanus Pre-conditioning; Test type: Other; p = 0.078, Log Rank

6. Secondary Outcome: Median Progression-free Survival in CMV Positive Participants
Description: Median progression-free survival will be estimated in the subset of participants that are CMV positive. Progression-free survival will be defined as the time in months between randomization and disease progression or death. Participants alive without disease progression will be censored at the time of their last follow-up. Kaplan-Meier methods will be used to estimate progression-free survival.
Time Frame: as for outcome 1
Population: Participants who are CMV positive. Data not collected on the Basiliximab and Tetanus pre-conditioning group.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group I: Unpulsed DC Pre-conditioning | Group II: Tetanus Pre-conditioning | Group III: Basiliximab and Tetanus Pre-conditioning
Number analyzed (Participants) | 9 | 11 | 0
months | 6.5 [4.4 to NA] — An estimation was not possible due to an insufficient number of participants experiencing events. | 6.8 [6.5 to NA] — An estimation was not possible due to an insufficient number of participants experiencing events. |
Statistical Analysis 1: Comparison: Group I: Unpulsed DC Pre-conditioning vs Group II: Tetanus Pre-conditioning; Test type: Other; p = 0.64, Log Rank

7. Secondary Outcome: Median Progression-free Survival in CMV Negative Participants
Description: Median progression-free survival will be estimated in the subset of participants that are CMV negative. Progression-free survival will be defined as the time in months between randomization and disease progression or death. Participants alive without disease progression will be censored at the time of their last follow-up. Kaplan-Meier methods will be used to estimate progression-free survival.
Time Frame: as for outcome 1
Population: Participants who are CMV negative. Data not collected on the Basiliximab and Tetanus pre-conditioning group.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group I: Unpulsed DC Pre-conditioning | Group II: Tetanus Pre-conditioning | Group III: Basiliximab and Tetanus Pre-conditioning
Number analyzed (Participants) | 16 | 16 | 0
months | 5.9 [4.1 to 14.7] | 5.8 [4.1 to 24.4] |
Statistical Analysis 1: Comparison: Group I: Unpulsed DC Pre-conditioning vs Group II: Tetanus Pre-conditioning; Test type: Other; p = 0.29, Log Rank

ADVERSE EVENTS:
Time Frame: Approximately 72 months (from the time of randomization of the first patient until approximately 31 months after randomization of the last patient)
Arm/Group | Group I: Unpulsed DC Pre-conditioning | Group II: Tetanus Pre-conditioning | Group III: Basiliximab and Tetanus Pre-conditioning
All-Cause Mortality (participants affected / at risk) | 24/27 | 22/28 | 6/9
Serious Adverse Events (participants affected / at risk) | 1/27 | 4/28 | 2/9
Other Adverse Events (participants affected / at risk) | 25/27 | 27/28 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group I: Unpulsed DC Pre-conditioning (N=27) | Group II: Tetanus Pre-conditioning (N=28) | Group III: Basiliximab and Tetanus Pre-conditioning (N=9)
Colonic perforation (Gastrointestinal disorders) | 0 | 0 | 1
Lung infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dysphasia (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Pyramidal tract syndrome (Nervous system disorders) | 0 | 1 | 1
Seizure (Nervous system disorders) | 0 | 2 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group I: Unpulsed DC Pre-conditioning (N=27) | Group II: Tetanus Pre-conditioning (N=28) | Group III: Basiliximab and Tetanus Pre-conditioning (N=9)
Anemia (Blood and lymphatic system disorders) | 13 | 15 | 6
Blood and lymphatic system disorders - Other, Specify (SWOLLEN LYMPH NODES BILATERAL NECK) (Blood and lymphatic system disorders) | 0 | 0 | 1
Chest pain - cardiac (Cardiac disorders) | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0
Blurred vision (Eye disorders) | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 2 | 0
Eye disorders - Other, Specify (DIFFICULTY WITH DEPTH PERCEPTION) (Eye disorders) | 0 | 0 | 1
Eye disorders - Other, Specify (L EYE REDNESS, INFLAMMATION) (Eye disorders) | 0 | 1 | 0
Eye disorders - Other, Specify (PERIPHERAL VISION LOSS) (Eye disorders) | 0 | 1 | 0
Floaters (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 4 | 2 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1
Fecal incontinence (Gastrointestinal disorders) | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 4 | 5 | 2
Vomiting (Gastrointestinal disorders) | 3 | 2 | 1
Edema face (General disorders) | 1 | 0 | 0
Edema limbs (General disorders) | 0 | 2 | 1
Fatigue (General disorders) | 2 | 4 | 2
Fever (General disorders) | 0 | 1 | 0
Flu like symptoms (General disorders) | 0 | 1 | 0
Gait disturbance (General disorders) | 1 | 1 | 0
Other, Specify (36 HOURS POST VACCINES, INCREASED CONFUSION, INCREASED FATIGUE, INCREASED APHASIA) (General disorders) | 0 | 1 | 0
Other, Specify (INTERMITTENT PULSATING IN EARS; POSSIBLE TINNITUS) (General disorders) | 0 | 1 | 0
Infusion related reaction (General disorders) | 0 | 1 | 1
Injection site reaction (General disorders) | 0 | 4 | 2
Localized edema (General disorders) | 0 | 0 | 1
Pain (General disorders) | 2 | 3 | 1
Allergic reaction (Immune system disorders) | 1 | 1 | 0
Bronchial infection (Infections and infestations) | 1 | 1 | 0
Infections and infestations - Other, Specify (BLEPHARITIS) (Infections and infestations) | 1 | 0 | 0
Infections and infestations - Other, Specify (ENLARGED AREAS UNDER ARMPITS) (Infections and infestations) | 1 | 0 | 0
Infections and infestations - Other, Specify (ORAL THRUSH) (Infections and infestations) | 0 | 1 | 0
Infections and infestations - Other, Specify (SHINGLES) (Infections and infestations) | 1 | 0 | 0
Infections and infestations - Other, Specify (TICK BITES) (Infections and infestations) | 1 | 0 | 0
Infections and infestations - Other, Specify (YEAST INFECTION) (Infections and infestations) | 0 | 1 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 3 | 3
Upper respiratory infection (Infections and infestations) | 3 | 6 | 3
Urinary tract infection (Infections and infestations) | 1 | 2 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 3 | 0
Injury, poisoning and procedural complications - Other, Specify (CHIPPED TOOTH) (Injury, poisoning and procedural complications) | 0 | 1 | 0
Injury, poisoning and procedural complications - Other, Specify (DOG BITE) (Injury, poisoning and procedural complications) | 0 | 1 | 0
Injury, poisoning and procedural complications - Other, Specify (HEAD INJURY) (Injury, poisoning and procedural complications) | 0 | 1 | 0
Injury, poisoning and procedural complications - Other, Specify (L ELBOW INJURY FALLING OUT OF BED) (Injury, poisoning and procedural complications) | 0 | 0 | 1
Injury, poisoning and procedural complications - Other, Specify (LEFT SHIN WOUND) (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 4 | 2
Alkaline phosphatase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 3 | 3
Blood bilirubin increased (Investigations) | 1 | 3 | 0
CD4 lymphocytes decreased (Investigations) | 3 | 2 | 5
Creatinine increased (Investigations) | 4 | 3 | 2
Lymphocyte count decreased (Investigations) | 15 | 16 | 6
Neutrophil count decreased (Investigations) | 10 | 10 | 4
Platelet count decreased (Investigations) | 14 | 15 | 6
Weight loss (Investigations) | 0 | 1 | 0
White blood cell decreased (Investigations) | 11 | 12 | 4
Anorexia (Metabolism and nutrition disorders) | 2 | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 1
Glucose intolerance (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 14 | 14 | 6
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 2 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 1 | 3 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 1 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 8 | 4
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 6 | 2
Hypokalemia (Metabolism and nutrition disorders) | 4 | 4 | 2
Hyponatremia (Metabolism and nutrition disorders) | 2 | 5 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Musculoskeletal and connective tissue disorder - Other, Specify (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 3 | 3 | 1
Dysgeusia (Nervous system disorders) | 0 | 2 | 0
Dysphasia (Nervous system disorders) | 6 | 5 | 0
Facial muscle weakness (Nervous system disorders) | 0 | 1 | 1
Facial nerve disorder (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 4 | 1
Hydrocephalus (Nervous system disorders) | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 1 | 5 | 2
Movements involuntary (Nervous system disorders) | 0 | 0 | 2
Nervous system disorders - Other, Specify (FEELING OF HEAD SPINNING) (Nervous system disorders) | 1 | 0 | 0
Nervous system disorders - Other, Specify (LEFT HAND LIMP) (Nervous system disorders) | 1 | 0 | 0
Nervous system disorders - Other, Specify (RESTLESSNESS) (Nervous system disorders) | 0 | 1 | 0
Nervous system disorders - Other, Specify (RIGHT ARM SENSATION) (Nervous system disorders) | 0 | 1 | 0
Nervous system disorders - Other, Specify (VISUAL FIELD CUT - HEMIANOPSIA) (Nervous system disorders) | 0 | 1 | 0
Paresthesia (Nervous system disorders) | 1 | 1 | 2
Presyncope (Nervous system disorders) | 0 | 1 | 0
Pyramidal tract syndrome (Nervous system disorders) | 0 | 1 | 1
Seizure (Nervous system disorders) | 7 | 8 | 2
Spasticity (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 2 | 0
Confusion (Psychiatric disorders) | 0 | 2 | 1
Insomnia (Psychiatric disorders) | 1 | 2 | 1
Hematuria (Renal and urinary disorders) | 1 | 1 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 3 | 2
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Skin and subcutaneous tissue disorders - Other, Specify (NIGHT SWEATS) (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, Specify (PIMPLE LIKE AREA NEAR SITE OF INJECTION) (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin and subcutaneous tissue disorders - Other, Specify (RASH) (Skin and subcutaneous tissue disorders) | 2 | 3 | 4
Skin and subcutaneous tissue disorders - Other, Specify (SKIN "SORENESS" AROUND L EYE) (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 22 | 24 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-20): https://cdn.clinicaltrials.gov/large-docs/28/NCT02366728/Prot_SAP_000.pdf